CLINICAL TRIAL: NCT07408037
Title: Preoperative Anxiety and Postoperative Recovery Delirium Observation in Children Who Underwent Gamified Breathing Exercise
Brief Title: Preoperative Gamified Breathing Exercise on Anxiety and Delirium in Children.
Acronym: PED-ANX-DEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Gulay Oztas, Research Assistant, PhD Student, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023-28 / 20
Record Dates: First submitted 2026-01-25; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Preoperative Anxiety (Ameliyat Öncesi Anksiyete); Emergence Delirium (Derlenme Deliryumu); Postoperative Complications; Pediatric Patients
Keywords: Preoperative Anxiety; Emergence Delirium; Gamification; Breathing Exercises; Pediatric Nursing; Postoperative Recovery
MeSH Terms: conditions — Emergence Delirium; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: A randomized controlled, parallel-group trial design is used to compare the effects of preoperative gamified breathing exercises with routine care. Participants are assigned to either the intervention group or the control group using a randomization method with numbered cards. Both groups receive the same baseline measurements, but only the intervention group undergoes the gamified breathing exercise protocol before surgery.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The primary and secondary outcomes (anxiety and delirium scores) are assessed by a blinded assistant researcher and a recovery room nurse who are unaware of the group assignments (intervention vs. control). This ensures that the evaluation of the Modified Yale Preoperative Anxiety Scale (mYPAS-SF) and the Pediatric Anesthesia Emergence Delirium (PAED) scale is conducted without bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified Breathing Exercise Group (Experimental): Participants in this group receive preoperative training on gamified breathing exercises. The intervention includes various interactive breathing games such as ball blowing, bubble blowing, candle blowing, or using breathing apps. Children are asked to perform these exercises for 10 minutes every hour, approximately 10-15 times per day, from 48-72 hours before surgery until the day of the operation.
  Interventions: Behavioral: Gamified Breathing Exercises
- No Intervention (No Intervention): his group receives routine preoperative information and standard care only. No gamified breathing exercises are practiced by the participants in this group.

INTERVENTIONS:
Behavioral: Gamified Breathing Exercises — The intervention involves providing preoperative training to children and their parents on gamified breathing exercises starting 48-72 hours before surgery. Children choose from various interactive breathing games, including:
  Ball Blowing: Blowing cotton or ping-pong balls across a surface using a straw.
  Bubble Blowing: Blowing soap bubbles to promote slow, deep exhalation.
  Candle Blowing: Practicing controlled breathing by blowing out candles.
  Tissue/Paper Blowing: Using breath to lift tissues or move paper windmills.
  Participants are instructed to practice these games for 10 minutes every hour, approximately 10-15 times per day, until the day of surgery. All necessary equipment (straws, bubbles, toys) is provided by the researchers.
  Arms: Gamified Breathing Exercise Group

SUMMARY:
This study aims to evaluate the effect of preoperative gamified breathing exercises on preoperative anxiety and postoperative emergence delirium in children. The intervention includes games like ball blowing and bubble blowing. Anxiety is measured using the mYPAS-SF scale, and delirium is assessed with the PAED scale.

DETAILED DESCRIPTION:
This randomized controlled study investigates the impact of preoperative gamified breathing exercises on preoperative anxiety and postoperative emergence delirium in pediatric patients. Children in the intervention group and their parents receive specialized training on gamified breathing exercises starting 48-72 hours before surgery.

The intervention consists of various interactive breathing games selected based on the child's preference, including:

Ball Blowing: Blowing a cotton or ping-pong ball across a flat surface or into a 'goal' using a straw to encourage deep exhalation.

Bubble Blowing: Using soap bubbles to promote slow and controlled breathing patterns.

Tissue/Paper Blowing: Blowing on tissues to lift them or move paper windmills.

Candle Blowing: Simulating or practicing blowing out candles using different breath strengths.

Participants are asked to perform these exercises for 10 minutes every hour, approximately 10-15 times per day, until the time of surgery. The control group receives routine preoperative information and care.

Primary outcomes are measured using the Modified Yale Preoperative Anxiety Scale (mYPAS-SF) before the operation. Postoperative emergence delirium is assessed in the recovery room at 0, 15, and 30 minutes using the Pediatric Anesthesia Emergence Delirium (PAED) scale."

Bu Bölümden Sonraki Adım: Arms and Interventions Bu metni kaydedip ilerlediğinizde, sistem sizden grupları (Arms) ve müdahaleleri (Interventions) ayrı ayrı tanımlamanızı isteyecektir.

Arm 1 (Experimental): Gamified Breathing Exercise Group.

Arm 2 (No Intervention/Control): Routine Care Group.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 7 years (preschool age).

Scheduled for elective (planned) surgery at Bursa Uludag University Hospital.

Physical status classified as ASA I or ASA II.

Children and parents who volunteer to participate and provide written informed consent.

Exclusion Criteria:

Children with chronic neurological or psychiatric disorders.

Children with existing respiratory system diseases that prevent breathing exercises.

Children or parents with communication barriers (e.g., severe hearing or speech impairment).

Children undergoing emergency (non-elective) surgery.

-

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2026-11-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Preoperative Anxiety Score | Immediately before the surgery (preoperative holding area).
  This will be assessed using the Modified Yale Preoperative Anxiety Scale-Short Form (mYPAS-SF). The scale evaluates five categories of behavior: activity, vocalization, emotional expressivity, state of arousal, and use of parents. Scores range from 22.92 to 100, where higher scores indicate higher levels of anxiety.

SECONDARY OUTCOMES:
Postoperative Emergence Delirium Level | At 0, 15, and 30 minutes after arrival in the Post-Anesthesia Care Unit (PACU).
  This will be assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale. The scale consists of five items: eye contact, purposeful actions, awareness of surroundings, restlessness, and inconsolability. Scores range from 0 to 20, with a score of 10 or higher indicating the presence of emergence delirium.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludağ Üniversitesi Hastanesi, Bursa, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] King-Underwood L, Pritchard-Jones K. Wilms' tumor (WT1) gene mutations occur mainly in acute myeloid leukemia and may confer drug resistance. Blood. 1998 Apr 15;91(8):2961-8. PMID 9531607
- [Result] Ebrahim GJ. The urban child's health and environment. J Trop Pediatr. 1997 Oct;43(5):253-4. doi: 10.1093/tropej/43.5.253. No abstract available. PMID 9364121
- [Result] Barreto Filho JB, Eiras PR, Golgher RR. N-terminal amino acids of bovine alpha interferons are relevant for the neutralization of their antiviral activity. Braz J Med Biol Res. 2001 May;34(5):663-7. doi: 10.1590/s0100-879x2001000500015. PMID 11323754